CLINICAL TRIAL: NCT02594501
Title: COBRA PzF Stenting to Reduce the Duration of Triple Therapy in Patients Treated With Oral Anticoagulation Undergoing Percutaneous Coronary Intervention
Brief Title: Randomized Trial of COBRA PzF Stenting to Reduce Duration of Triple Therapy
Acronym: COBRA-REDUCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: CeloNova BioSciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COBRA 2015-01
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Angina, Stable; Angina, Unstable; Anticoagulants
MeSH Terms: conditions — Angina, Stable; Angina, Unstable | interventions — Drug-Eluting Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- COBRA PzF (Experimental): Cobra PzF plus 14-day DAPT (dual antiplatelet therapy)
  Interventions: Device: COBRA PzF
- Drug Eluting Stent (Active Comparator): standard FDA-approved DES (Xience/Promus or Resolute) plus 3 or 6-month DAPT (dual anti-platelet therapy)
  Interventions: Device: Drug Eluting Stent

INTERVENTIONS:
Device: COBRA PzF
  Arms: COBRA PzF
Device: Drug Eluting Stent
  Other Names: Xience/Promus, Resolute or Synergy
  Arms: Drug Eluting Stent

SUMMARY:
The purpose of this study is to determine whether patients undergoing coronary intervention that also require oral anticoagulation, treatment with the COBRA PzF stent plus 14-day dual anti-platelet therapy (DAPT) has higher safety and non-inferior outcomes for thrombo-embolic events than compared with standard FDA-approved drug eluting stent (DES) plus 3 or 6-month DAPT.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than age 18 with ischemic symptoms (stable or unstable angina or NSTEMI without thrombosis of the target lesion on coronary angiography) or evidence of myocardial ischemia in the presence of ≥ 50% de novo stenosis located in native coronary vessels (max. 2 lesions in one or 2 separate vessels).
* Patient receiving or with an indication for new treatment with long-term oral anticoagulation with a coumadin derivatives or non-vitamin K oral anticoagulants.
* Written, informed consent

Exclusion Criteria:

* Cardiogenic shock
* Target lesion located in left main trunk
* Bifurcation interventions with a planned 2-stent strategy
* Vessel size too small for implantation of a 2.5 mm stent by visual estimation
* Patient requiring staging PCI procedure within 6 months after the index procedure
* Patients requiring DAPT for more than 2 weeks after the index procedure
* Contraindications or allergy to cobalt, chromium, platinum, polyzene-F, everolimus, zotarolimus or the inability to take triple therapy for at least 6 months
* Relevant hematologic deviations: platelet count <100x10^9 cells/L or >600x10^9 cells/L
* Active bleeding; bleeding diathesis; recent trauma or major surgery in the last month; history of intracranial bleeding or structural abnormalities; suspected aortic dissection
* Malignancies or other co-morbid conditions with life expectancy less than 12 months or that may result in protocol non-compliance
* Pregnancy, present (positive pregnancy test), suspected or planned, breast feeding
* Known allergy or intolerance to the study medications: ASA, clopidogrel, coumadin and its derivatives
* Patient's inability to fully cooperate with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 996 (Actual)
Dates: Start 2016-02-05; Primary Completion 2021-05 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
BARC class >=2 bleeding after hospital discharge (or beyond 14 days, whichever is "later"). | 6 months
Composite of all cause death, myocardial infarction, definite and probable stent thrombosis or ischemic stroke | 6 months

SECONDARY OUTCOMES:
Composite of all cause death, myocardial infarction, definite and probable stent thrombosis, ischemia-driven target lesion revascularization or ischemic stroke | 12 months
Composite of cardiac death and myocardial infarction | 12 months
Ischemia driven target lesion revascularization | 12 months
Definite and probable stent thrombosis | 12 months
Ischemic stroke | 12 months
BARC class 3-5 bleeding | 6 months
TIMI major bleeding; TIMI major and minor bleeding | 6 months
Acute Success Rates | procedure
  Device success; Lesion success; Procedure success
Health economic utility | 12 months
  Total cardiovascular and bleeding related costs with cost effectiveness based on events avoided

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Kastrati, Study Chair — ISAResearch Center Deutsches Herzzentrum München
Locations (48):
- United States (22):
  - Christiana Care Health Services, Newark, Delaware
  - University of Florida, Jacksonville, Florida
  - Memorial Hospital Jacksonville, Jacksonville, Florida
  - Sebastian River Medical Center, Melbourne, Florida
  - Mt Sinai Medical Center, Miami Beach, Florida
  - Augusta University, Augusta, Georgia
  - University of Maryland St. Joseph Medical Center, Towson, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Rutgers Robert Wood Johnson Medical Schoo, New Brunswick, New Jersey
  - Northwell Health, Manhasset, New York
  - NYU Winthrop Hospital, Mineola, New York
  - North Ohio Heart Center, Elyria, Ohio
  - Cleveland Clinic, Fairview Park, Ohio
  - Mercy St. Vincent Medical Center, Toledo, Ohio
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - Texas Cardiac Center, Lubbock, Texas
  - Tyler Cardiovascular Consultants, Tyler, Texas
  - Sentara Heart Hospital (Sentara Cardiovascular Research Institute), Norfolk, Virginia
  - Carilion Medical Center, Roanoke, Virginia
  - Charleston Area Medical Center, Charleston, West Virginia
- ZNA Middelheim, Antwerp, Belgium
- Aarhus University Hospital, Aarhus, Denmark
- France (7):
  - Clinique Axium, Aix
  - Clinique Du Pont De Chaumes, Montauban
  - Clinique du Millénaire, Montpellier
  - Hopital Pitie-Salpitierre, Paris
  - Höpital George Pompidou, Paris
  - Clinique Pasteur, Toulouse
  - Institut Lorrain du Coeur et Vaisseaux, CHU Nancy-Barbois, Vandœuvre-lès-Nancy
- Germany (13):
  - Universitats Herzzentrum Freibourg, Bad Krozingen
  - Charité - Campus Benjamin Franklin, Berlin
  - Uni-Klinikum Erlangen, Erlangen
  - St. Josefskrankenhaus, Freiburg im Breisgau
  - Klinikum Fürth, Fürth
  - University of Jena, Jena
  - MediClin Herzzentrum, Lahr
  - Klinikum Landshut-Achdorf, Landshut
  - Deutsches Herzzentrum München, Munich
  - Klinikum Rechts der Isar München, Munich
  - Universitätsklinikum Regensburg, Regensburg
  - Hegau Bodensee Klinikum Singen, Singen
  - Univesitätsklinikum Tübingen, Tübingen
- Ospedale Spaziani, Frosinone, Italy
- Paula Stradins Clinical University Hospital, Riga, Latvia
- Switzerland (2):
  - Hopital Cantonal Fribourg, Fribourg
  - Kantonspital St Galen, Sankt Gallen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byrne RA, Colleran R, Coughlan JJ, Jauhar R, Maillard L, De Labriolle A, Maeng M, Croft C, Brunner M, Leistner D, Zrenner B, Kollum M, Laugwitz KL, Xhepa E, Mayer K, Lahu S, Joner M, Kirtane A, Mehran R, Barakat M, Urban P, Cutlip DE, Kastrati A; COBRA-REDUCE Investigators. Randomized Trial of COBRA PzF Stenting to Reduce the Duration of Triple Therapy: The COBRA-REDUCE Trial. Circ Cardiovasc Interv. 2024 Oct;17(10):e013735. doi: 10.1161/CIRCINTERVENTIONS.123.013735. Epub 2024 Oct 15. PMID 39405373
- [Derived] Colleran R, Joner M, Cutlip D, Urban P, Maeng M, Jauhar R, Barakat M, Michel JM, Mehran R, Kirtane AJ, Maillard L, Kastrati A, Byrne RA; COBRA-REDUCE investigators. Design and Rationale of a Randomized Trial of COBRA PzF Stenting to REDUCE Duration of Triple Therapy (COBRA-REDUCE). Cardiovasc Revasc Med. 2022 Jan;34:17-24. doi: 10.1016/j.carrev.2021.01.022. Epub 2021 Jan 22. PMID 33608239